CLINICAL TRIAL: NCT02649517
Title: Clinical and Morphological Characteristics of Chronic Inflammation in the Myocardium in Patients With Decompensated Heart Failure With Ischemic Systolic Dysfunction
Brief Title: Clinical and Morphological Characteristics of Chronic Inflammation in the Myocardium in Patients With Decompensated HF With Ischemic Systolic Dysfunction
Acronym: FHID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Vyacheslav Ryabov, MD,PhD Research Institute for Cardiology, Russian Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1801
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Decompensated Heart Failure; Ischemic Heart Disease
Keywords: decompensated heart failure; ischemic heart disease; inflammatory cardiomyopathy
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- chronic inflammation (Other): All patients will be held PCI to exclude ischemic heart failure decompensation. Also, all patients will be performed endomyocardial biopsy.
  Interventions: Procedure: Endomyocardial biopsy

INTERVENTIONS:
Procedure: Endomyocardial biopsy — Endomyocardial biopsy will be performed through a puncture in the femoral vein. 3-6 samples taken under the control of myocardial echocardiography or flyuroskopii. Samples of biopsy material then transmitted Pathomorphology for immunohistochemistry, light microscope.
  Other Names: EMB

SUMMARY:
The purpose of the study is to investigate the clinical and morphological characteristics of chronic subclinical inflammation in the myocardium in patients with decompensated heart failure with ischemic systolic dysfunction.

DETAILED DESCRIPTION:
Important reason for the development of chronic heart failure is a viral disease of the heart, the three phenotypes associated with: the presence of inflammation without viral agent, implying an autoimmune disease; presence of inflammation and persistent viruses; and the presence of persistent virus without signs of inflammation.

There is a group of patients with coronary heart disease, which on the background of optimal treatment is observed progression of clinical symptoms of coronary heart disease with the subsequent development of heart failure, leading to ischemic cardiomyopathy. Perhaps the reason for this is the combination of inflammatory and ischemic cardiomyopathies.

Inflammatory cardiomyopathy, involved in the pathogenesis of DCM, includes idiopathic, autoimmune and infectious subtypes. Inflammatory disease of the myocardium diagnosed by established histological, immunological and immunohistochemical criteria.

This study will include 60 patients with decompensated heart failure with ischemic left ventricular systolic dysfunction (LVEF <40%) were hospitalized not earlier than 6 months after myocardial revascularization. This group of patients will receive standard treatment, according to national guidelines RSC and ESC, to stabilize heart failure. All patients will be held PCI to exclude ischemic heart failure decompensation. Also, all patients will be performed endomyocardial biopsy as a result of immunohistochemical studies will be made on the separation of the virus and the virus-negative-positive group. After that, the group will be divided into subgroups: virus - and inflammation in the myocardium inflammation without viral antigen, viral inflammation of the presence of antigen and the group with the presence of viral antigen without any signs of inflammation in the myocardium.

The study is nonrandomized.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over the age of 18 years old and weighing up to 130 kg
* Clinical symptoms of decompensated heart failure in history
* Heart failure decompensation requiring hospitalization for at least 3 of the following symptoms: shortness of breath, or position orthopnea, rales, peripheral edema, jugular venous pulsations, signs of stagnation in the pulmonary circulation according to the X-ray of the chest
* Confirmed coronary heart disease with diastolic dysfunction (LVEF <40%) in history and at the time of admission
* The term of the inclusion of patients in the study did not earlier than six months after revascularization (PCI or CABG)
* Patients receiving medical treatment according to national guidelines RSC and ESC with individually tailored doses of drugs

Exclusion Criteria:

* The refusal of a patient to conduct the necessary studies
* Poor visualization of the heart when ultrasound
* Hemodynamically significant valvular heart disease
* Acute coronary syndrome
* Тhrombosis of the right atrium and right ventricle
* Condition after the operation, impeding access to the right ventricle (cava filters plication vena cava, Mustard or Senning operation on the d-transposition of the great arteries, a mechanical prosthetic tricuspid valve)
* Severe comorbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of inflammatory infiltrate in the myocardial tissue | 6 month after PCI or CABG

SECONDARY OUTCOMES:
Incidence of the virus - positive inflammatory infiltrate in the myocardial tissue | 6 month after PCI or CABG
The most frequent viral agents in myocardial tissue in this region | 6 month after PCI or CABG
Incidence of the acute myocardial infarction | 6 and 12 month after PCI or CABG
Incidence of disturbance rhythm and conduction of the heart | 6 and 12 month after PCI or CABG
Left ventricular ejection fraction (Echo) | 6 and 12 month after PCI or CABG
Еnd-diastolic volume of the left ventricle (Echo) | 6 and 12 month after PCI or CABG
Еnd-systolic volume of the left ventricle (Echo) | 6 and 12 month after PCI or CABG
Incidence of the mortality | 6 and 12 month after PCI or CABG
Incidence of the stroke | 6 and 12 month after PCI or CABG
Incidence of hospitalizations for decompensation heart failure | 6 and 12 month after PCI or CABG

CONTACTS AND LOCATIONS:
Overall Officials: Vyacheslav Ryabov, MD, PhD, Principal Investigator — Research Institute for Cardiology
Locations (2):
- Russia (2):
  - Research Institutite for Cardiology, Tomsk, Tomskii Region
  - Scientific and Research Institution of Cardiology of Siberian Department of RAMS, Tomsk